CLINICAL TRIAL: NCT02881528
Title: Autoimmune Diabetes Accelerator Prevention Trial - adAPT Stage 1
Brief Title: Autoimmune Diabetes Accelerator Prevention Trial
Acronym: adAPT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor Recruitment prior to end of funding timelines.
Sponsor: University of Exeter (Other)
Collaborators: University of Dundee (Other); University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15/135763; 2015-000748-41 (EudraCT Number); 15/ES/0075 (Other: Research Ethics Committee)
Record Dates: First submitted 2016-03-28; First posted 2016-08-29 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Prediabetic State
Keywords: Type 1 Diabetes; Juvenile Diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 1 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin Hydrochloride (Experimental): Metformin Hydrochloride Ph Eur oral solution (100mg/1ml) Starting Dose 10mg/Kg body weight once daily for 2 weeks, increasing to 10mg/Kg body weight twice daily if tolerated, increasing to target dose of 20mg/Kg body weight twice daily (max 1000mg twice daily) at Month 1 (4 weeks post randomization).
  Down-titration to 10mg/kg twice daily if target dose not tolerated. Stage 1: Dosing for up to 15 months (option to extend to Stage 2: 36 months)
  Interventions: Drug: Metformin Hydrochloride
- Placebo (Placebo Comparator): Placebo (100mg/1ml) Starting Dose 10mg/Kg body weight once daily for 2 weeks, increasing to 10mg/Kg body weight twice daily if tolerated, increasing to target dose of 20mg/Kg body weight twice daily (max 1000mg twice daily) at Month 1 (4 weeks post randomization).
  Down-titration to 10mg/kg twice daily if target dose not tolerated. Stage 1: Dosing for up to 15 months (option to extend to Stage 2: 36 months)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — Liquid formula metformin administered by oral syringe in a dose of 10mg/kg body weight once daily for 2 weeks, then to 10mg/Kg twice daily (maximum 500mg twice daily) for a further two weeks during the first month, increasing to 20mg/kg body weight twice daily (maximum 1000mg twice daily) thereafter.
  Other Names: Metformin
  Arms: Metformin Hydrochloride
Drug: Placebo — Liquid formula of placebo administered by oral syringe in an equivalent volume to a metformin dose of 10mg/kg body weight once daily for 2 weeks, then to 10mg/Kg twice daily (maximum 500mg twice daily) for a further two weeks during the first month, increasing to 20mg/kg body weight twice daily (maximum 1000mg twice daily) thereafter.
  Arms: Placebo

SUMMARY:
The autoimmune diabetes ACCELERATOR PREVENTION TRIAL (adAPT) is based on the accelerator hypothesis. The trial is designed to establish whether metformin, an oral hypoglycaemic agent that is known to reduce insulin demand in type 2 diabetes (T2D), can do the same in children at risk of type 1 diabetes (T1D) and thereby prevent disease.

The first phase of adAPT will screen participants aged 5-16 years (inclusive) for islet-related autoantibodies who are the siblings or offspring of individuals diagnosed with T1D before the age of 25years in Scotland and England.

There are four principle islet-related antibodies associated with T1D. The presence of two or more confers a 40% risk of developing T1D in five years. While the presence of none or one antibody carries a similar risk for developing T1D to the general population (1 in 500 in 5years).

It is anticipated that 5% of those screened will be identified as double-antibody positive, these participants will be invited to join the intervention phase of the study - randomised controlled trial (RCT). Up to 200 eligible subjects could be identified by screening with a minimum of 90 being enrolled into the RCT phase.

adAPT is a proposed three stage project. The current protocol defines the screening phase, Stage 1 and seamless entry into Stage 2. Screening will identify children and young people at high risk of developing T1D and invite them to participate in Stage 1 which will involve a minimum of 4 months treatment with either metformin/placebo, however Stage1 treatment will run seamlessly into Stage 2. Stage 1/2 treatment will last up to 21 months (to accommodate 15months screening, 4 months treatment and 2 months analysis). Post Stage1 analysis/ late Stage 2 participation will last up to 36 months (participants enrolled early into Stage 1 will have the longest intervention).

During the Stage1 participants will be tested on three occasions (baseline, month 1 and month 4) for metabolic response using a 5-point mixed meal tolerance test (MMTT). Testing will continue in Stage 1/2 with 3 visits further visits at months 8, 12, 18. Late Stage 2 visits will occur on months 24, 30 & 36.

Participants will be invited to continue into Stage 3, taking treatment up to 60 months post analysis of Stage 1 and associated protocol amendment and additional consent.

DETAILED DESCRIPTION:
adAPT is a randomised double-blind placebo-controlled Phase IV clinical trial.

Metformin, a licensed medicine but will be tested out with its current license (off-label). Participants will either receive metformin (liquid) or matched placebo in a double blind manner; neither the participant or study team will know the allocation.

Metformin, the study medication, reduces the demand for insulin in Type 2 diabetes (T2D). adAPT will test if metformin can also reduce insulin demand in children at risk of Type 1 Diabetes (T1D). adAPT has an adaptive design with each stage informing the next with progression depend upon the previous stages outcome Stage 1 exposes each participant to metformin or placebo for four months, following which they seamlessly enter Stage 2. However, because recruitment rolls over 15 months many of those recruited early on will have entered Stage 2 before some even reach Stage 1. Accordingly, the protocol and submission also outlines Stages 2.

A successful Stage 1 will lead-on to a clinical outcome trial (Stages 2 and 3) which, if successful, will fundamentally change our understanding of what causes diabetes and how to prevent it. Stage 1 is required to confirm that adAPT trial design is achievable. Outcome evaluation will be undertaken at 21 months. Stage 2 (proof-of-concept) will test if metformin can slow-down the development of diabetes. The outcome data form Stage 1 will allow for power to be calculated to drive the number of participants required for the study for Stages 2 (and 3). It is proposed that once the power and thus population numbers are established for Stage 2 (out with this protocol) that new participants will enter Stage 1 via screening and follow the established trial pathway.

Diabetes biological markers will be measured and formally assessed at the end of Stage 2, after 36 months. Stage 3 will occur if metformin treatment in Stage 2 is proven to be better than placebo for slowing the development of diabetes. Stage 3 will further investigate the development of diabetes between the groups, using biological markers and clinical outcomes at five years.

Children/adolescents aged between 5-16 years (inclusive) at the time of screening and who are siblings or offspring of people diagnosed with type 1 diabetes before the age of 25 are eligible to be invited to participate in the screening phase of adAPT. Families/ children will be invited to participate in screening and will informed of the study by invitation letter (via the index T1D patient) from their designated clinician/Principal Investigator (PI) or via their family practitioner through Scottish Primary Care Research Network/Clinical Research Network (SPCRN/CRN). In addition potential participants may contact the study team independently (self-referral) in response to media/press and internet coverage. Those invited via letter will be requested to either return the reply slip, or call/Short Message Service (SMS)/email the study team to register their interest.

Parent and child age-appropriate Screening Information will be provided and written consent and assent will be completed. Consent/assent will only occur after a minimum of 24 hours has elapsed from study information provision.

Screening will take place in clinically appropriate locations. Screening requires a small non-fasting blood sample (3.5 mls). Participants will be offered topical anaesthesia prior to the blood sample being taken.

This sample will be tested for four islet-related antibodies. Two or more antibodies will infer a positive test, while one or less will conclude a negative test. It is anticipated that approximately 5% of the screened population will present with a positive results and thus a 40% risk of diabetes over 5 years and thus are eligible to be invited into Stage 1 of the study. It is expected that 95% of people screened will test negative and their participation will conclude (except for remote data linkage relating to diabetes diagnosis for 10 years post study participation). The antibody tests are posted to the study's partner laboratory in Bristol, United Kingdom (UK) with results being available within an 8 week timeframe.

Antibody positive participants/families will receive a result consultation and an invitation to the intervention stage of the study. Age-appropriate information sheets will be provided for children/adolescents in addition to parents/guardian information.

If child/adolescent and parent/guardian assent/consent to participant in the RCT phase the following visits will take place:

Stage 1 Month 0 (M0) visit - lasting approximately 2.5 to 3 hours:

Measure participant height, weight and waist circumference. Urine pregnancy test for all menstruating female participants. Topical anaesthesia will be offered and applied if participant agreeable. (Following assessment of anaesthesia) a cannula will be inserted for blood sampling.

Safety blood samples to measure fasting glucose levels, full blood count, liver function, urea and electrolytes. Samples sent to local National Health Service (NHS) hospital accredited laboratories.

Research blood samples: Antibodies, Immunology, deoxyribonucleic acid (DNA -with consent and Vitamin B12.

Mixed Meal Tolerance Testing (MMTT) baseline samples (Insulin, C-peptide and Glucose) followed by Ensure Plus (or equivalent) drink at 6ml per kg dose (maximum 360ml) with 4 further blood tests being obtained at 30 minute intervals (via the in situ cannula) for 2 hours; Time points: 0, 30, 60, 90, 120 minutes.

Randomisation will occur following eligibility criteria and safety sample results review by PI. If the participant is not eligible the participant and parent will be informed of the rationale for non-eligibility and the participant' s family doctor will be informed of any clinically significant findings (with consent.) Participants will be provided with study medication (Metformin or placebo) and given instructions on dose and administration after randomisation has taken place at M0 visit.

If eligible, more than one sibling can be screened and, if seropositive, recruited. To avoid treatment contamination, immediate family members will be allocated to the same treatment group, with the first family member tested being the one who is randomly allocated.

The required study medication dose is calculated using the participant's weight using a dosing algorithm using 2.5kg increments to the nearest 0.5mls.

On commencement of treatment metformin can cause gastric intolerance, therefore to minimise side effects for the first two weeks participants will be requested to take once daily 10mg/kg - half the target dose. Medication is administered/ taken orally.

Month 0 + 2 weeks:

Research nurse will contact the parent/participant to review tolerability and if tolerated increase to twice daily dosing of 10mg/kg and will assess adverse event profile. New written dosing instructions will be provided. If the participant is not tolerating dose they will be withdrawn from the study.

Month 1 Visit - lasting approximately 2.5 to 3 hours:

Procedures are the same as M0 without an antibody blood sample. Study medication is increased to the target dose of 20mg/kg, twice daily. Participants are provided with new written dosing instructions.

Month 1 + 1 week:

Research nurse will phone the parent/participant to review tolerability of up-titrated dose and assess adverse event profile. If the dose is not tolerated they their dose will be reduced to the previous tolerated dose of 10mg/kg, twice a day which will continue for the remainder of the trial. Where down-titration occurs new written dosing instructions will be provided.

Month 4, 8, 12, 18, (Late Stage 2: 24, 30, 36) - lasting approximately 2.5 to 3 hours:

Procedures are the same as M0 with antibody sample. Clinical significant results will reported as per local laboratory ranges and protocol.

Months 1, 2 & 3 and every 3 months or as required the research nurse will contact parent/participant to assess adverse event profile.

ELIGIBILITY:
Inclusion Criteria -For Screening

* Aged 5-16years (inclusive) at time of screening
* Offspring of parents or siblings who themselves developed T1D before the age of 25years
* Parent /Participant is willing and able to give informed consent/assent

Additional Inclusion Criteria for Intervention Phase

• Individuals identified by screening to be sero-positive for at least two of the four islet-related antibodies; Insulin Autoantibodies (IAA), Islet Antigen-2 Autoantibodies (IA-2A), Glutamic Acid Decarboxylase Autoantibodies (GADA), Zinc Transporter 8 Autoantibodies (ZnT8).

Exclusion Criteria for Screening:

* Parent /Participant is unwilling/unable to give informed consent/assent
* Under 5y or over 17y at time of screening
* Offspring of parents or siblings who themselves developed T1D after the age of 25years
* Known to have physician diagnosed diabetes
* Already taking metformin
* Physically or psychologically unable to participate
* Taking medication likely to increase insulin resistance or blood glucose levels (e.g. oral/systemic; steroids, growth hormone, beta-2-agonists, diuretics or angiotensin-converting-enzyme (ACE) -inhibitors.)
* Suffering from anoxia, cardiovascular insufficiency, renal or hepatic disease or sepsis - contraindication to metformin
* Participating in another clinical trial (other than observational trials and registries) concurrently or within 30 days prior to screening for entry into this study

Additional Exclusion Criteria for Intervention Phase:

* Development of diabetes during the screening phase
* Identified by screening to be sero-negative (fewer than two of the four islet-related antibodies (IAA, GAD, IA-2, ZnT8)
* Fasting Blood Glucose of ≥ 7 mmol/L at Month 0
* Postmenarche female participants of childbearing potential who are pregnant or lactating
* Postmenarche female participants of childbearing potential must be sexually abstinent or use another acceptable form of contraception during study participation
* Renal failure or renal dysfunction (creatinine clearance < 60 mL/min)
* Acute conditions with the potential to alter renal function such as, severe infection, shock
* Acute or chronic disease which may cause tissue hypoxia such as: cardiac or respiratory failure, recent myocardial infarction, shock, hepatic insufficiency acute alcohol intoxication, alcoholism
* Known allergies to milk and/or soya
* Hypersensitivity to metformin hydrochloride or any of the excipients: Parahydroxybenzoates may cause allergic reactions (possibly delayed); Liquid mannitol - patients with rare hereditary fructose intolerance.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Between group difference in reduction of Homeostatic Model Assessment (HOMAR) of Insulin Resistance (IR, mass units). | 21 months (Stage1)
  Note: study not powered to nominate a primary outcome as feasibility study.
Between group difference in reduction in beta cell demand as measured by serum glucose (mmol/L) and C-peptide (ng/mL) | 21 months
  Note: study not powered to nominate a primary outcome as feasibility study.

SECONDARY OUTCOMES:
Feasibility of a randomized controlled trial in children who are at high risk of T1D as measured by recruitment rates (%) | 21 months
Feasibility of a randomized controlled trial in children who are at high risk of T1D as measured by attrition rates (%) | 21 months

OTHER OUTCOMES:
Percentage response rate of families who choose to participate in the intervention stage when a second sibling in the same family is found to be at high risk of T1D. | 21 months
  Calculate the response rate of those identified as double antigen positive and decide to participate in the RCT phase of the study.
Compliance with study medication. | 21 months (Stage1)
  Adherence measured as a percentage of prescribed doses.
Between group difference in serum vitamin B12 | 21 months (Stage1)
Between group difference in Immunological t-cell response to diabetes | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Rob Andrews, Prof, Principal Investigator — University of Exeter
Locations (5):
- United Kingdom (5):
  - NHS Ayrshire & Arran, Kilmarnock, Ayrshire
  - NHS Grampian, Aberdeen, Grampian
  - NHS Lanarkshire, Wishaw, Lanarkshire
  - NHS Tayside, Dundee, Tayside
  - NHS Greater Glasgow & Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: No